CLINICAL TRIAL: NCT05613322
Title: Resistell Phenotech AST to Determine the Antibiotic Susceptibility of Gram-negative Bacteria Causing Bacteremia: a Prospective, Non-interventional, Multi-centric, Clinical Performance Study
Brief Title: Resistell Phenotech AST to Determine the Antibiotic Susceptibility of Gram-negative Bacteria Causing Bacteremia
Acronym: PHENOTECH-1
Status: Terminated | Type: Observational
Why Stopped: Statistical power for primary endpoint (sensitivity) for E. coli and K. pneumoniae and ceftriaxone was achieved
Sponsor: Resistell AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PHENOTECH-1
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Bacteremia Sepsis
Keywords: Antibiotic; Susceptibility; AST; E.coli; K. pneumoniae; Phenotech
MeSH Terms: conditions — Disease Susceptibility; Escherichia coli Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacteria extracted from blood and tested with the investigational device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Resistell Phenotech — Resistell Phenotech IVD device used to assess susceptibility of Gram negative bacteria to antibiotics.

SUMMARY:
The aim of this study is to assess the sensitivity, specificity, and accuracy of the Resistell Phenotech device in testing antibiotic susceptibility of Gram-negative bacteria (i.e., E. coli or K. pneumoniae) to clinically relevant antibiotics. The study is designed as a prospective, non-interventional, multi-center, single-arm study.

The blood culture samples from bacteremia patients that are positive for E. coli or K. pneumoniae will be tested with the Resistell Phenotech device after strain identification by MALDI-TOF. The results of the Resistell AST will be compared with the results from the disk diffusion tests (all sites use the Kirby-Bauer disk diffusion test), and site dependent tests (VITEK® 2, BD Phoenix™, MicroScan WalkAway system, and/or EUCAST RAST), which are currently the standard AST methods in the microbiology laboratories at the participating sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed a General Consent form approving use of their residual blood samples for research purposes (applicable at CHUV only)
* Patients who have signed a consent allowing the use of their residual sample (Restprobenerklärung) (applicable at MUI, only)
* Patients over the age of 18 years (>18)
* Patients with bacteremia considered to be due to E. coli or K. pneumoniae
* Patients whose positive blood cultures were not older than 24 hours at the time of AST start

Exclusion Criteria:

* Patients with documented refusal of the use of biological material for research purposes (applicable at CHUV, only)
* Patients with polymicrobial bacteremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bacteremia considered to be due to E. coli or K. pneumoniae.
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the Resistell Phenotech vs Kirby-Bauer | 18 months
  To assess the sensitivity of the Resistell Phenotech in detecting antibiotic susceptible bacteria in blood samples positive for E. coli or K. pneumoniae, compared to the gold standard Kirby-Bauer disk diffusion test.

SECONDARY OUTCOMES:
Specificity and accuracy of the Resistell Phenotech vs Kirby-Bauer | 18 months
  To assess the specificity and accuracy of the Resistell Phenotech in detecting antibiotic susceptible bacteria in blood samples positive for E. coli or K. pneumoniae, compared to the gold standard Kirby-Bauer disk diffusion test.
Sensitivity, specificity, and accuracy of the Resistell Phenotech vs other comparators | 18 months
  To assess the sensitivity, specificity, and accuracy of the Resistell Phenotech in detecting antibiotic susceptible bacteria in blood samples positive for E. coli or K. pneumoniae, compared to other routine diagnostic AST tests run at each site
Time to result of Resistell Phenotech vs Kirby-Bauer and other comparators | 18 months
  To assess the difference between time to result (TTR) of Resistell Phenotech and the TTR of the Kirby-Bauer and the other routine diagnostic AST methods run at each site.
Category agreement and discrepancies | 18 months
  To assess category agreement (CA), very major discrepancy (VMD), major discrepancy (MD) of the results obtained with Resistell Phenotech compared to the Kirby-Bauer and the other routine diagnostic AST test results at each site

CONTACTS AND LOCATIONS:
Locations (3):
- Medizinische Universität Innsbruck (MUI), Institut für Hygiene und Medizinische Mikrobiologie, Innsbruck, Innsbruck, Austria
- Hospital Universitario Ramón y Cajal, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Madrid, Spain
- Centre hospitalier universitaire vaudois (CHUV), Institut de Microbiologie, Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided